CLINICAL TRIAL: NCT03369769
Title: Physiological Wellness Effects of Animal-assisted Activities in Children With Autism Spectrum Disorder in a Specialized Psychiatric Hospital Program
Brief Title: Wellness Effects of Animal-assisted Activities With Autism Spectrum Disorder Youth in a Specialized Psychiatric Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Human Animal Bond Institute for Research (Unknown); Purdue University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-1227
Record Dates: First submitted 2017-10-24; First posted 2017-12-12 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Child Behavior; Autism Spectrum Disorder; Psychiatric Hospitalization; Veterinary Therapeutics
MeSH Terms: conditions — Child Behavior; Autism Spectrum Disorder | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: To investigate the effect of canine animal assisted activities (AAA) on physiological arousal levels in children and adolescents with autism spectrum disorder (ASD) (ages 4 to 17 years) in a specialized psychiatric hospital program. It is hypothesized that children with ASD will demonstrate lower physiological arousal in the presence of canines, compared to a non-animal control.
Who Masked: Outcomes Assessor
Masking Description: Coders for the videotaped behavioral data collected via the OHAIRE-M tool were blind to specific study objective.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canine & Adult Handler Activity (Experimental): Unstructured 10-minute small group interaction with canine & handler
  Interventions: Other: Activity
- Toy and Adult Handler Activity (Active Comparator): Unstructured 10-minute small group interaction with toy & handler
  Interventions: Other: Activity

INTERVENTIONS:
Other: Activity — 10 minutes interaction with therapy dog and adult handler in small group (2-4 participants).
  Other Names: animal-assisted activity (AAA)

SUMMARY:
Background: Children with Autism Spectrum Disorder (ASD) are at higher risk for developing co-existing mental health conditions and consequently experiencing psychiatric hospitalization, compared to the general pediatric population. However, hospital environments can be exceptionally stressful for this population, given their social-communication deficits, ineffective emotional regulation skills and heightened physiological arousal. While the use of animal-assisted activities (AAA) show potential for various improvements in children with ASD in community settings, these "stress-reducing" and "social-buffering" benefits have not yet been studied within a psychiatric hospital setting for youth with ASD.

Objectives: Evaluate whether an AAA with canines can lead to reduced physiological arousal and improvements in social-communication as well as aberrant behaviors in children and adolescents diagnosed with ASD in a specialized psychiatric hospital setting.

Methods: Participants were recruited from the Neuropsychiatric Special Care (NSC) program's inpatient and/or partial day-treatment program. Prior to study participation, baseline demographic measures were acquired from caregivers and participants' ASD diagnosis was confirmed. Participants experienced two, randomly assigned 35-minute sessions (AAA and Control Condition) with a minimum two-day washout period between groups. Each session included a baseline 20-minute social skills group immediately followed by a 10 minute experimental or control condition. The AAA condition introduced a canine and volunteer handler for free interaction time while the control condition introduced a novel toy and a volunteer for free interaction. Participants' physiological arousal was continuously assessed throughout all conditions via the Empatica E-4 wristbands (Empatica Inc. 2014). All sessions were videotaped for behavioral coding using the Observation of Human Animal Interaction for Research - Modified, v.1.

DETAILED DESCRIPTION:
Background: Children with ASD are at higher risk for developing co-existing mental health conditions and consequently experiencing psychiatric hospitalization, compared to the general pediatric population. However, hospital environments can be exceptionally stressful for this population, given their social-communication deficits, ineffective emotional regulation skills and heightened physiological arousal. While the use of animal-assisted activities (AAA) show potential for various improvements in children with ASD in community settings, these "stress-reducing" and "social-buffering" benefits have not yet been studied within a psychiatric hospital setting for youth with ASD.

Objectives: Evaluate whether an AAA with canines can lead to reduced physiological arousal and improvements in social-communication as well as aberrant behaviors in children and adolescents diagnosed with ASD in a specialized psychiatric hospital setting.

Methods: Participants were recruited from the Neuropsychiatric Special Care (NSC) program's inpatient and/or partial day-treatment program. Prior to study participation, baseline demographic measures were acquired from caregivers and participants' ASD diagnosis was confirmed. Participants experienced two, randomly assigned 35-minute sessions (AAA and Control Condition) with a minimum two-day washout period between groups. Each session included a baseline 20-minute social skills group immediately followed by a 10 minute experimental or control condition. The AAA condition introduced a canine and volunteer handler for free interaction time while the control condition introduced a novel toy and a volunteer for free interaction. Participants' physiological arousal was continuously assessed throughout all conditions via the Empatica E-4 wristbands (Empatica Inc. 2014). All sessions were videotaped for behavioral coding using the Observation of Human Animal Interaction for Research - Modified, v.1.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a specialized psychiatric unit for children with developmental disabilities
* Meeting standard cut-off scores for ASD on the Social Communication Questionnaire Screener (> 12) and Autism Diagnostic Observation Schedule-2nd Ed
* English speaking

Exclusion Criteria:

* Unwillingness to wear wristband & be videotaped
* Allergies or phobias to canines
* Inability to attend to and participate in a social group
* Prisoner status or ward of the state

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Change in physiological measurements with the wristband device from baseline through 90 minutes. | Baseline; 90 minutes
  The Wristband device is worn by the participant for 90 minutes during the day of the experimental condition. Physiological measure of Galvanic skin response, heart rate, heart rate variability will be assessed at baseline through 90 minutes. Collection points during this day includes comparison from baseline, social group, and experimental condition.

SECONDARY OUTCOMES:
Observation of Human Animal Interaction for Research (OHAIRE-modified) | Two 10-minute conditions (experimental and control) on two separate days.
  The Observation of Human-Animal Interaction for Research (OHAIRE) is a timed interval coding system intended to capture the unique interactions between humans and animals. It was originally developed and piloted with children with autism spectrum disorder (ASD) interacting with typically-developing peers in a small group school setting with guinea pigs compared to toys.

CONTACTS AND LOCATIONS:
Overall Officials: Robin L Gabriels, Psy.D., Principal Investigator — University of Colorado, Denver

REFERENCES:
- [Background] Germone MM, Gabriels RL, Guerin NA, Pan Z, Banks T, O'Haire ME. Animal-assisted activity improves social behaviors in psychiatrically hospitalized youth with autism. Autism. 2019 Oct;23(7):1740-1751. doi: 10.1177/1362361319827411. Epub 2019 Feb 28. PMID 30818971